CLINICAL TRIAL: NCT02284594
Title: Adult Influenza Vaccination Text Message Reminders With Electronic Health Record Alerts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Assistant Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAK5058_3
Record Dates: First submitted 2014-11-03; First posted 2014-11-06 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- text message (Experimental): Receipt of series of text messages regarding influenza vaccination
  Interventions: Behavioral: text message
- usual care (No Intervention)

INTERVENTIONS:
Behavioral: text message — series of text messages regarding influenza vaccination
  Arms: text message

SUMMARY:
Influenza infection leads to on average 3000-49,0000 deaths and 150,000 hospitalizations annually. While vaccination is the cornerstone of preventing influenza infection, vaccination coverage in adults is low. Latino adults have the lowest coverage rates. Text message reminders have been used successfully for improving influenza vaccination for children. This study will assess the use of text messaging to improve influenza vaccination coverage rates in a largely minority, publicly insured adult population. We will also assess if the patient having received a text message makes the patient more likely to accept vaccination when their provider has received in electronic alert regarding need for influenza vaccination in the electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years of age
* at least one visit to the AIM clinic during previous 6 months
* a cell phone number in the registration system
* fluent in English or Spanish

Exclusion Criteria:

- Receipt of influenza vaccination during the 2014-2015 influenza season prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4026 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
influenza vaccination | up to 5 months
  receipt of influenza vaccine

SECONDARY OUTCOMES:
influenza vaccination | up to 2 months
  receipt of influenza vaccine
captured opportunity | up to 5 months
  receipt of influenza vaccination during a visit

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center/ NewYork Presbyterian Hospital Ambulatory Care Network, New York, New York, United States